CLINICAL TRIAL: NCT07394101
Title: Pharmacokinetic Characterization of Tartaric Acid in Humans: Effect of the Food Matrix (Wine, Grapes, and Juice) on Its Bioavailability
Brief Title: Pharmacokinetic Characterization of Tartaric Acid in Humans
Acronym: TARBIO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anallely Lopez, Postdoctoral Researcher, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HCB/2025/1296
Record Dates: First submitted 2026-02-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Adult Participants; Non-smoking, Healthy Adults; Normal Weight Adults
Keywords: Tartaric acid; Pharmacokinetics; Bioavailability; Food matrix effect; Wine; Healthy volunteers
MeSH Terms: interventions — Wine; whole grape extract

STUDY DESIGN:
Intervention Model Description: This is a randomized, partially blinded, interventional study designed to evaluate the effects of different polyphenol-containing matrices on healthy adults. Thirty healthy non-smoking participants (aged 20-40 years, BMI 23-27 kg/m²), without a history of cardiovascular, hepatic, or renal disease, and not following any special diet for at least 4 weeks prior to the study, will be recruited. Participants will be randomly assigned to one of three intervention groups (wine, grape, or juice) using a block randomization system stratified by sex to ensure a 1:1 balance across groups. The study will be partially blinded: participants will be unaware of the study hypothesis, but not the intervention, due to the nature of the matrices.
Masking Description: Masking will be partial: participants will be blind to hypotheses but not to the intervention (due to the nature of the matrices).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Red Wine (Experimental): Participants will consume 100 mL of red wine, providing a standardized dose of tartaric acid, after a 10-hour overnight fast. The wine will be ingested within 5 minutes, accompanied by a standardized meal (2 slices of white bread) to simulate real-life consumption conditions. Intake of other fluids will be controlled (water ad libitum except during the first hour), and compliance will be monitored through direct observation.
  Interventions: Dietary Supplement: Wine
- Grape fruits (Experimental): Participants will consume a portion of fresh grapes containing an equivalent dose of tartaric acid to the wine, following the same controlled conditions: after a 10-hour overnight fast, ingested within 5 minutes with the standardized meal, with controlled fluid intake and direct compliance monitoring.
  Interventions: Dietary Supplement: Grape
- Grape juice (Experimental): Participants will consume 150 mL of grape juice standardized for tartaric acid content, under identical conditions: after a 10-hour overnight fast, ingested within 5 minutes with the standardized meal, with controlled fluid intake and compliance monitoring.
  Interventions: Dietary Supplement: Juice

INTERVENTIONS:
Dietary Supplement: Wine — 100 mL of red wine containing a standardized dose of tartaric acid, ingested after a 10-hour overnight fast with a standardized meal (2 slices of white bread). Consumption completed within 5 minutes, fluid intake controlled, compliance monitored.
  Arms: Red Wine
Dietary Supplement: Grape — Portion of fresh grapes providing an equivalent dose of tartaric acid as the wine, consumed under the same controlled conditions.
  Arms: Grape fruits
Dietary Supplement: Juice — 150 mL of grape juice standardized for tartaric acid content, ingested under identical conditions as the other arms.
  Arms: Grape juice

SUMMARY:
The goal of this clinical trial is to characterize the pharmacokinetics (absorption, distribution, metabolism, and excretion; ADME) and oral bioavailability of tartaric acid in humans after its administration through different food matrices (red wine, fresh grapes, and grape juice). The study aims to determine whether the pharmacokinetic behavior of tartaric acid is matrix-dependent and dose-dependent in healthy adult volunteers.

The main questions it aims to answer are:

Does the food matrix (wine, grapes, or grape juice) influence the oral bioavailability of tartaric acid?

Are there differences in key pharmacokinetic parameters of tartaric acid, including maximum plasma concentration (Cmax), time to reach maximum concentration (Tmax), total exposure (AUC), half-life (t1/2), and urinary excretion, depending on the matrix of intake?

Researchers will compare the pharmacokinetic profiles of tartaric acid after consumption in red wine, grapes, and grape juice to evaluate differences in absorption, systemic exposure, and elimination attributable to the source of intake.

Participants will:

Follow a polyphenol-restricted diet prior to the study, including avoidance of grapes, wine, and related products.

Consume a single standardized dose of tartaric acid administered as red wine, fresh grapes, or grape juice after an overnight fast.

Provide blood samples at multiple time points over a 24-hour period to determine plasma tartaric acid concentrations.

Collect urine samples over 24 hours for assessment of tartaric acid excretion.

Consume standardized low-polyphenol meals under controlled conditions during the study day.

DETAILED DESCRIPTION:
This study will characterize the pharmacokinetics (absorption, distribution, metabolism, and excretion) and oral bioavailability of tartaric acid (TA) in humans after consumption in different food matrices: red wine, fresh grapes, and grape juice. Although moderate wine consumption has been associated with cardiometabolic benefits, the human pharmacokinetics of TA-the main organic acid in grapes and wine-remain largely uncharacterized. Existing data from animal studies do not account for the influence of the food matrix on absorption or systemic exposure.

TA has been proposed as an objective biomarker of wine intake, and its dietary presence may contribute to observed cardiovascular and anti-inflammatory effects. Bioavailability of bioactive compounds is strongly matrix-dependent, and interactions within complex foods can enhance or limit absorption. This study provides the first direct evaluation of whether TA pharmacokinetics differ depending on the food matrix.

Using a randomized, parallel-group design, participants will receive a standardized dose of TA in one of the three matrices, with plasma and urine samples analyzed by advanced LC-MS/MS methods. Results will establish reference pharmacokinetic parameters, clarify the effect of the food matrix on TA bioavailability, and support development of functional grape-derived products, while improving interpretation of epidemiological evidence linking TA to cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking adults aged 20-40 years.
* Body mass index (BMI) between 23 and 27 kg/m².
* No history of cardiovascular, hepatic, or renal disease.
* No adherence to any special diet for at least 4 weeks prior to the study.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Current smokers or recent ex-smokers.
* History of cardiovascular, hepatic, or renal disorders.
* Current adherence to any special diet or nutritional supplementation that could affect study outcomes.
* Any condition or medication that could interfere with absorption, metabolism, or excretion of tartaric acid.
* Participation in another clinical trial within the past 3 months.
* Pregnancy or lactation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Oral bioavailability of tartaric acid | 0-24 hours post-ingestion
  Quantification of the oral bioavailability of tartaric acid after administration in different dietary matrices (wine, grape, grape juice) using dose-response studies.
Maximum plasma concentration (Cmax) | 0-24 hours, sampling at 0, 15, 30 min, 1, 2, 3, 4, 6, 8, and 24 h post-ingestion
  Determination of the peak plasma concentration of tartaric acid in human plasma using liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS).
Time to reach maximum plasma concentration (Tmax) | 0-24 hours, sampling at 0, 15, 30 min, 1, 2, 3, 4, 6, 8, and 24 h post-ingestion
  Time required to reach the Cmax of tartaric acid in plasma.
Area under the plasma concentration-time curve (AUC) | 0-24 hours, sampling at 0, 15, 30 min, 1, 2, 3, 4, 6, 8, and 24 h post-ingestion
  Total plasma exposure of tartaric acid determined by non-compartmental analysis using WinNonlin.

SECONDARY OUTCOMES:
Plasma half-life (t1/2) | 0-24 hours, sampling at 0, 15, 30 min, 1, 2, 3, 4, 6, 8, and 24 h post-ingestion
  Time required to reduce plasma tartaric acid concentration by half, calculated using non-compartmental analysis.
Maximum cumulative urinary concentration | 0-24 hours, collected in fractions: 0-4, 4-8, 8-12, and 12-24 h post-ingestion
  Maximum amount of tartaric acid excreted in urine, measured by LC-ESI-MS/MS.
Comparison of pharmacokinetic parameters by matrix | grape, grape juice) to assess matrix- and dose-dependence. 0-24 hours post-ingestion
  Comparison of Cmax, Tmax, AUC, and t1/2 between dietary matrices (wine, grape, grape juice) to assess matrix- and dose-dependence.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Hospital Clínic, Institut d'Investigació Biomèdica August Pi i Sunyer, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No